CLINICAL TRIAL: NCT04884763
Title: A Randomized, Double Blind, Placebo-Controlled Single Center Phase 2 Pilot Study to Assess the Safety and Efficacy of Off-label Subcutaneous Administration of Erenumab-aooe in Patients With Temporomandibular Disorder
Brief Title: Safety and Efficacy of Erenumab-aooe in Patients With Temporomandibular Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: Amgen (Industry)
Responsible Party: Principal Investigator, Domenick Zero, Professor, Department of Biomedical and Applied Sciences, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20-D-242; CAMG334AUS01T (Other: Novartis Investigator Initiated Trials (IITs) Program)
Record Dates: First submitted 2021-05-04; First posted 2021-05-13 (Actual); Results first posted 2025-08-19 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-07

CONDITIONS: Temporomandibular Disorder
MeSH Terms: conditions — Temporomandibular Joint Disorders | interventions — erenumab

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A (Active Comparator): Arm A: erenumab-aooe (EREN) 140 mg s.c. administered every four weeks for a total of five treatments
  Interventions: Drug: Erenumab-aooe (EREN) 140 mg s.c. administered every four weeks for a total of five treatments
- Arm B (Placebo Comparator): Arm B: placebo (EREN-P) s.c. administered every four weeks for a total of five treatments
  Interventions: Drug: Placebo (EREN-P) s.c. administered every four weeks for a total of five treatments

INTERVENTIONS:
Drug: Erenumab-aooe (EREN) 140 mg s.c. administered every four weeks for a total of five treatments — Erenumab-aooe (EREN) 140 mg s.c. administered at baseline and weeks 4, 8, 12 and 16 for a total of five treatments
  Other Names: Aimovig®
  Arms: Arm A
Drug: Placebo (EREN-P) s.c. administered every four weeks for a total of five treatments — Placebo (EREN-P) s.c. administered at baseline and weeks 4, 8, 12 and 16 for a total of five treatments
  Other Names: Placebo
  Arms: Arm B

SUMMARY:
The purpose of this proof of concept study is to evaluate the safety and efficacy of the off-label use of Aimovig® (EREN) in reducing Temporomandibular Disorder (TMD) pain compared to placebo.

DETAILED DESCRIPTION:
This will be a 24-week, randomized, double-blinded, placebo-controlled, parallel group proof-of-concept study with two arms (active and placebo). The plan is to enroll 30 subjects. There will be a four-week screening period to identify subjects that meet the diagnostic criteria (DC/TMD) for "myalgia", recommended by the International RDC/TMD Consortium Network and Orofacial Pain Special Interest Group. The Diagnostic Criteria for Temporomandibular Disorders Symptom Questionnaire and DC/TMD Examination Form will be used during Screening and Baseline visits to confirm the TMD diagnosis and determine whether subjects meet the inclusion/exclusion criteria.

Subjects will attend a Screening visit followed by Baseline visit to randomize eligible subjects to active (EREN) or placebo (EREN-P). During the Baseline visit and Wks 4, 8, 12, and 16, subjects will receive treatment with either 140 mg of EREN or Placebo administered by subcutaneous injection. At Baseline and Wks 4, 8, 12, 16, 20, and 24 subjects will be instructed to complete the Brief Pain Inventory (BPI); PEG (Pain, Enjoyment, General Activity) Scale; pain mediation assessment; Patient Global Impression of Change (PGIC) (except for Baseline visit); Jaw Function Limitation Scale (JFLS); Patient Health Questionnaire (PHQ-4); and Somatic Symptom Scale (SSS-8). These visits will include review of continuance criteria and adverse event collection.

At the Screening and Baseline visits the subjects will be instructed on how to use the PEG Scale and pain use assessment app, which will be downloaded on their smartphone, to provide a daily assessment of their pain intensity and interference with enjoyment and general activity (PEG) and their daily used of pain medications. Subjects who do not own a smartphone or are unwilling to use the app on a daily basis will only complete the PEG and pain medication assessment at the Baseline visit and all subsequent visits using the app onsite.

ELIGIBILITY:
Inclusion Criteria:

Subjects eligible for inclusion in the study must meet all of the following criteria:

1. Signed the informed consent;
2. Have pain-related TMD myalgia assessed by history and clinical examination as established by the DC/TMD;
3. Age 18 years and younger than 60 years;
4. Have a good knowledge of the English language;
5. Able to understand and comply with the study requirements;
6. Have had TMD myalgia for 6 months or longer; and
7. If taking pain medications, the dose regimen must be stable for at least 4 weeks prior to the screening visit.

Exclusion Criteria:

Subjects meeting any of the following criteria are not eligible for inclusion:

1. Lacking stable bilateral posterior occlusion;
2. Currently uses a complete maxillary or mandibular prosthetic denture;
3. Currently pregnant or plan to become pregnant;
4. Breastfeeding or plan to breastfeed;
5. Allergic to erenumab-aooe or any of the ingredients in Aimovig® (acetate, polysorbate 80, and sucrose);
6. Allergic to rubber or latex;
7. Currently undergoing TMD treatment elsewhere;
8. Currently undergoing orthodontic treatment;
9. Currently included in other experimental protocols within the last 30 days before enrollment;
10. Having 11 or more headaches during the past 4 weeks;
11. Having received massage, acupuncture or physical therapy treatment of the head, neck or shoulders during the previous 3 months;
12. History of unstable or acute severe pain from another pain condition;
13. History of traumatic brain injury;
14. History of surgical treatment or recommended surgical treatment for TMD;
15. History of ongoing, unresolved disability litigation;
16. History of drug abuse;
17. History of moderate to severe sleep apnea requiring CPAP or oral mandibular repositioning appliance;
18. Anything that would place the subjects at increased risk or preclude the individual's full compliance with or completion of the study (e.g., medical condition, laboratory finding, physical exam finding logistical complication); and
19. History of previously receiving erenumab-aooe or other anti-CGRP therapies, including anti-CGRP and anti-CGRP receptor monoclonal antibodies and small molecule CGRP receptor antagonists (gepants).
20. History of chronic constipation and/or using medication associated with decreased gastrointestinal motility.
21. History of hypertension or risk factors for hypertension.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2021-11-15 (Actual); Primary Completion 2024-01-04 (Actual); Study Completion 2024-01-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Domenick T Zero, DDS, MS, Principal Investigator — Indiana University; Harold C Avila, DDS, MS, Principal Investigator — Indiana University; Kurt Kroenke, MD, MACP, Principal Investigator — Regenstrief Institute, Inc.
Locations (1):
- Indiana University School of Dentistry, Oral Health Research Institute, Indianapolis, Indiana, United States

REFERENCES:
- [Background] Ashina M, Goadsby PJ, Reuter U, Silberstein S, Dodick D, Rippon GA, Klatt J, Xue F, Chia V, Zhang F, Cheng S, Mikol DD. Long-term safety and tolerability of erenumab: Three-plus year results from a five-year open-label extension study in episodic migraine. Cephalalgia. 2019 Oct;39(11):1455-1464. doi: 10.1177/0333102419854082. Epub 2019 May 30. PMID 31146544
- [Background] de Leeuw, R, Editor, Orofacial Pain: Guidelines for Assessment, Diagnosis, and Management, The American Academy of Orofacial Pain, Sixth Edition, Hanover Park, IL: Quintessence Publishing Co, Inc., 2018, 1-2
- [Background] Edvinsson L. The CGRP Pathway in Migraine as a Viable Target for Therapies. Headache. 2018 May;58 Suppl 1:33-47. doi: 10.1111/head.13305. PMID 29697153
- [Background] Goadsby PJ, Reuter U, Hallstrom Y, Broessner G, Bonner JH, Zhang F, Sapra S, Picard H, Mikol DD, Lenz RA. A Controlled Trial of Erenumab for Episodic Migraine. N Engl J Med. 2017 Nov 30;377(22):2123-2132. doi: 10.1056/NEJMoa1705848. PMID 29171821
- [Background] Hargreaves R, Olesen J. Calcitonin Gene-Related Peptide Modulators - The History and Renaissance of a New Migraine Drug Class. Headache. 2019 Jun;59(6):951-970. doi: 10.1111/head.13510. Epub 2019 Apr 25. PMID 31020659
- [Background] Headache Classification Committee of the International Headache Society (IHS). The International Classification of Headache Disorders, 3rd edition (beta version). Cephalalgia. 2013 Jul;33(9):629-808. doi: 10.1177/0333102413485658. No abstract available. PMID 23771276
- [Background] Julious SA. Sample size of 12 per group rule of thumb for a pilot study. Pharmaceutical statistics. 2005;4:287-291.
- [Background] Kean J, Monahan PO, Kroenke K, Wu J, Yu Z, Stump TE, Krebs EE. Comparative Responsiveness of the PROMIS Pain Interference Short Forms, Brief Pain Inventory, PEG, and SF-36 Bodily Pain Subscale. Med Care. 2016 Apr;54(4):414-21. doi: 10.1097/MLR.0000000000000497. PMID 26807536
- [Background] Krebs EE, Lorenz KA, Bair MJ, Damush TM, Wu J, Sutherland JM, Asch SM, Kroenke K. Development and initial validation of the PEG, a three-item scale assessing pain intensity and interference. J Gen Intern Med. 2009 Jun;24(6):733-8. doi: 10.1007/s11606-009-0981-1. Epub 2009 May 6. PMID 19418100
- [Background] Kroenke K, Evans E, Weitlauf S, McCalley S, Porter B, Williams T, Baye F, Lourens SG, Matthias MS, Bair MJ. Comprehensive vs. Assisted Management of Mood and Pain Symptoms (CAMMPS) trial: Study design and sample characteristics. Contemp Clin Trials. 2018 Jan;64:179-187. doi: 10.1016/j.cct.2017.10.006. Epub 2017 Oct 12. PMID 29031492
- [Background] Kroenke K, Krebs EE, Turk D, Von Korff M, Bair MJ, Allen KD, Sandbrink F, Cheville AL, DeBar L, Lorenz KA, Kerns RD. Core Outcome Measures for Chronic Musculoskeletal Pain Research: Recommendations from a Veterans Health Administration Work Group. Pain Med. 2019 Aug 1;20(8):1500-1508. doi: 10.1093/pm/pny279. PMID 30615172
- [Background] Kroenke K, Spitzer RL, Williams JB, Lowe B. An ultra-brief screening scale for anxiety and depression: the PHQ-4. Psychosomatics. 2009 Nov-Dec;50(6):613-21. doi: 10.1176/appi.psy.50.6.613. PMID 19996233
- [Background] Maixner W, Fillingim RB, Williams DA, Smith SB, Slade GD. Overlapping Chronic Pain Conditions: Implications for Diagnosis and Classification. J Pain. 2016 Sep;17(9 Suppl):T93-T107. doi: 10.1016/j.jpain.2016.06.002. PMID 27586833
- [Background] Noseda R, Burstein R. Migraine pathophysiology: anatomy of the trigeminovascular pathway and associated neurological symptoms, cortical spreading depression, sensitization, and modulation of pain. Pain. 2013 Dec;154 Suppl 1:S44-53. doi: 10.1016/j.pain.2013.07.021. Epub 2013 Jul 25. PMID 23891892
- [Background] Ohrbach, R, editor. Diagnostic Criteria for Temporomandibular Disorders Assessment Instruments. Version 15May2016. www.rdc-tmdinternational.org Accessed on 23Sep2019
- [Background] Ohrbach R, Granger C, List T, Dworkin S. Preliminary development and validation of the Jaw Functional Limitation Scale. Community Dent Oral Epidemiol. 2008 Jun;36(3):228-36. doi: 10.1111/j.1600-0528.2007.00397.x. PMID 18474055
- [Background] Popko L. Some Notes on Papyrus Ebers, Ancient Egyptian Treatments of Migraine, and a Crocodile on the Patient's Head. Bull Hist Med. 2018;92(2):352-366. doi: 10.1353/bhm.2018.0030. PMID 29961718
- [Background] Schiffman E, Ohrbach R, Truelove E, Look J, Anderson G, Goulet JP, List T, Svensson P, Gonzalez Y, Lobbezoo F, Michelotti A, Brooks SL, Ceusters W, Drangsholt M, Ettlin D, Gaul C, Goldberg LJ, Haythornthwaite JA, Hollender L, Jensen R, John MT, De Laat A, de Leeuw R, Maixner W, van der Meulen M, Murray GM, Nixdorf DR, Palla S, Petersson A, Pionchon P, Smith B, Visscher CM, Zakrzewska J, Dworkin SF; International RDC/TMD Consortium Network, International association for Dental Research; Orofacial Pain Special Interest Group, International Association for the Study of Pain. Diagnostic Criteria for Temporomandibular Disorders (DC/TMD) for Clinical and Research Applications: recommendations of the International RDC/TMD Consortium Network* and Orofacial Pain Special Interest Groupdagger. J Oral Facial Pain Headache. 2014 Winter;28(1):6-27. doi: 10.11607/jop.1151. PMID 24482784
- [Background] Speciali JG, Dach F. Temporomandibular dysfunction and headache disorder. Headache. 2015 Feb;55 Suppl 1:72-83. doi: 10.1111/head.12515. Epub 2015 Feb 3. PMID 25644695
- [Background] Tepper SJ. History and Review of anti-Calcitonin Gene-Related Peptide (CGRP) Therapies: From Translational Research to Treatment. Headache. 2018 Nov;58 Suppl 3:238-275. doi: 10.1111/head.13379. Epub 2018 Sep 22. PMID 30242830
- [Background] Tepper S, Ashina M, Reuter U, Brandes JL, Dolezil D, Silberstein S, Winner P, Leonardi D, Mikol D, Lenz R. Safety and efficacy of erenumab for preventive treatment of chronic migraine: a randomised, double-blind, placebo-controlled phase 2 trial. Lancet Neurol. 2017 Jun;16(6):425-434. doi: 10.1016/S1474-4422(17)30083-2. Epub 2017 Apr 28. PMID 28460892
- [Background] Toussaint A, Kroenke K, Baye F, Lourens S. Comparing the Patient Health Questionnaire - 15 and the Somatic Symptom Scale - 8 as measures of somatic symptom burden. J Psychosom Res. 2017 Oct;101:44-50. doi: 10.1016/j.jpsychores.2017.08.002. Epub 2017 Aug 2. PMID 28867423
- [Background] Yuan H, Spare NM, Silberstein SD. Targeting CGRP for the Prevention of Migraine and Cluster Headache: A Narrative Review. Headache. 2019 Jul;59 Suppl 2:20-32. doi: 10.1111/head.13583. PMID 31291020
- [Derived] Avila HC, Kroenke K, Eckert GJ, Gossweiler AG, Galvez LDC, Zero DT. A randomized, double blind, placebo-controlled pilot study to assess the efficacy of erenumab in individuals with temporomandibular disorder. J Oral Facial Pain Headache. 2025 Jun;39(2):75-83. doi: 10.22514/jofph.2025.027. Epub 2025 Jun 12. PMID 41070535
- See also: Highlights of Prescribing Information — https://www.accessdata.fda.gov/drugsatfda_docs/label/2020/761077s007lbl.pdf

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm A | Arm B
Started | 15 | 15
4-week Visit | 12 | 15
8-week Visit | 12 | 15
12-week Visit | 11 | 13
16-week Visit | 11 | 13
20-week Visit | 9 | 12
24-week Visit | 10 | 12
Completed | 10 | 12
Not Completed | 5 | 3

BASELINE CHARACTERISTICS:
Population: Thirty-two patients met the inclusion/exclusion criteria. Two patients who qualified for the study were never randomized to study treatment; one decided not to continue and the other due to scheduling issues.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A | Arm B | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 15 | 15 | 30
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 34.9 [21 to 58] | 34.7 [23 to 52] | 34.8 [21 to 58]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 13 | 26
  Male | 2 | 2 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 3 | 8
  Not Hispanic or Latino | 9 | 12 | 21
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 14 | 14 | 28
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 15 | 15 | 30
Brief Pain Inventory (BPI) pain severity [Mean (Standard Deviation); unit: units on a scale] — Brief Pain Inventory (BPI) pain severity scale rates pain-related severity in 4 areas. Each item is rated on a 0 (no pain) to 10 (severe pain) scale. The BPI pain severity score is the average of the items and ranges from 0 (Better) - 10 (Worse).
  units on a scale | 3.0 (1.99) | 2.9 (1.35) | 2.95 (1.67)
Brief Pain Inventory (BPI) pain interference [Mean (Standard Deviation); unit: units on a scale] — Brief Pain Inventory (BPI) pain interference scale rates pain-related interference in 7 areas. Each item is rated on a 0 (does not interfere) to 10 (completely interferes) scale. The BPI pain interference score is the average of the items and ranges from 0 (Better) - 10 (Worse).
  units on a scale | 2.31 (1.90) | 2.07 (1.60) | 2.19 (1.73)
Pain Score [Mean (Standard Deviation); unit: units on a scale] — Pain score: 0 (Better) - 10 (Worse)
  units on a scale | 3.45 (2.54) | 3.62 (1.85) | 3.54 (2.15)
Jaw Function Limitation Scale (JFLS-8) [Mean (Standard Deviation); unit: units on a scale] — Jaw Function Limitation Scale (JFLS-8): 0 (Better) - 10 (Worse).
  units on a scale | 1.69 (1.21) | 1.81 (1.36) | 1.75 (1.27)
Patient Health Questionnaire (PHQ-4) [Mean (Standard Deviation); unit: units on a scale] — Patient Health Questionnaire (PHQ-4): 0 (Better) - 12 (Worse). Measure of depression and anxiety.
  units on a scale | 2.80 (2.54) | 2.27 (1.75) | 2.53 (2.16)
Somatic Symptoms Scale (SSS-8) [Mean (Standard Deviation); unit: units on a scale] — Somatic Symptoms Scale (SSS-8): 0 (Better) - 32 (Worse)
  units on a scale | 6.80 (4.81) | 8.60 (4.15) | 7.70 (4.51)

OUTCOME MEASURES:

1. Primary Outcome: Brief Pain Inventory (BPI) Pain Severity at 20 Weeks
Description: Assessment of pain severity using the Brief Pain Inventory (BPI) 4-item pain severity scale at 20 weeks: 0 (Better) - 10 (Worse). Interim assessments were performed at 4, 8, 12 and 16 weeks and post-treatment at 24 weeks (secondary outcome).
Time Frame: 20 weeks.
Population: Estimation done using mixed-model ANOVA which includes all available data from all time points for all subjects. This analysis reduces bias compared to an analysis at each time point that excludes subjects with missing data. All study subjects were included, even if they did not have data observed at the given time point. In addition to missing data shown in Participant Flow table, outcome-specific missing data for 1 additional Arm A subject at week 12 and 2 additional Arm B subjects at week 20.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 15 | 15
score on a scale | 1.72 [0.78 to 2.65] | 1.42 [0.55 to 2.29]
Statistical Analysis 1: Comparison: Arm A vs Arm B; Based on two-sided paired t-tests and two-sample t-tests, all conducted at a 5% significance level, this pilot study had 80% power to detect effect sizes of 1.2 for differences between groups. To account for dropout, the study enrolled 15 patients per group, for a total of 30 patients; Test type: Superiority; p = 0.567, Mixed Models Analysis — A two-sided 5% significance level was used for all tests without multiplicity adjustment between multiple endpoints; Model included factors for treatment group, time, and their interaction, with time repeated within subject. Gender as a covariate; Mean Difference (Final Values) = 0.30, 95% CI 2-sided [-0.76 to 1.35] — For difference calculation, Arm A - Arm B

2. Secondary Outcome: Brief Pain Inventory (BPI) Pain Interference at 20 Weeks
Description: Assessment of pain interference using the Brief Pain Inventory (BPI) 7-item pain intensity scale at 20 weeks: 0 (Better) - 10 (Worse). Interim assessments were performed at 4, 8, 12 and 16 weeks and post-treatment at 24 weeks (additional secondary outcome).
Time Frame: 20 weeks
Population: Estimation done using mixed-model ANOVA which includes all available data from all time points for all subjects. This analysis reduces bias compared to an analysis at each time point that excludes subjects with missing data. All study subjects were included, even if they did not have data observed at the given time point. In addition to missing data shown in Participant Flow table, outcome-specific missing data for 1 additional Arm A subject at week 12 and 1 additional Arm B subjects at week 20.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 15 | 15
score on a scale | 1.11 [0.28 to 1.94] | 0.96 [0.18 to 1.74]
Statistical Analysis 1: Comparison: Arm A vs Arm B; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.778, Mixed Models Analysis — A two-sided 5% significance level was used for all tests without multiplicity adjustment between multiple endpoints; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.15, 95% CI 2-sided [-0.91 to 1.21] — For difference calculation, Arm A - Arm B

3. Secondary Outcome: Average Daily Reported Pain Scores at 20 Weeks
Description: Assessment of pain using average of daily reported pain scores at 20 weeks; average of daily reported scores from days > week 16 and <= week 20. Pain scale: 0 (Better) - 10 (Worse). Interim assessments were performed at 4, 8, 12 and 16 weeks and post-treatment at 24 weeks (additional secondary outcome).
Time Frame: 20 weeks
Population: Estimation done using mixed-model ANOVA which includes all available data from all time points for all subjects. This analysis reduces bias compared to an analysis at each time point that excludes subjects with missing data. All study subjects were included, even if they did not have data observed at the given time point. In addition to missing data shown in Participant Flow table, outcome-specific missing data for 4 Arm A subjects at wk 0, 1 Arm A at wk 4, 1 Arm A at wk 12, and 2 Arm B at wk 0.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 15 | 15
score on a scale | 1.92 [0.94 to 2.90] | 1.04 [0.13 to 1.94]
Statistical Analysis 1: Comparison: Arm A vs Arm B; Based on two-sided paired t-tests and two-sample t-tests, all conducted at a 5% significance level, this pilot study had 80% power to detect effect sizes of 0.9 for changes over time within groups and effect sizes of 1.2 for differences between groups. To account for dropout, the study enrolled 15 patients per group, for a total of 30 patients; Test type: Superiority; p = 0.105, Mixed Models Analysis — A two-sided 5% significance level was used for all tests without multiplicity adjustment between multiple endpoints; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.88, 95% CI 2-sided [-0.20 to 1.96] — For difference calculation, Arm A - Arm B

4. Secondary Outcome: % of Days Taking Medication for Pain at 20 Weeks
Description: Assessment of pain using the % of days taking medication for pain at 20 weeks; percentage of days calculated from days > week 16 and <= week 20.Interim assessments were performed at 4, 8, 12 and 16 weeks and post-treatment at 24 weeks (additional secondary outcome).
Time Frame: 20 weeks
Population: Estimation done using mixed-model ANOVA which includes all available data from all time points for all subjects. This analysis reduces bias compared to an analysis at each time point that excludes subjects with missing data. All study subjects were included, even if they did not have data observed at the given time point. In addition to missing data shown in Participant Flow table, outcome-specific missing data for 1 additional Arm A subject at week 4 and 1 additional Arm A subject at week 12.
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage of days
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 15 | 15
percentage of days | 23.0 [0.8 to 45.1] | 5.4 [-14.4 to 25.2]
Statistical Analysis 1: Comparison: Arm A vs Arm B; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.163, Mixed Models Analysis — A two-sided 5% significance level was used for all tests without multiplicity adjustment between multiple endpoints; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 17.5, 95% CI 2-sided [-7.6 to 42.7] — For difference calculation, Arm A - Arm B

5. Secondary Outcome: Pain Improvement Using the Patient Global Impression of Change in Pain at 20 Weeks
Description: Assessment of pain improvement using the patient global impression of change in pain scale at 20 weeks: 1 (Better) - 7 (Worse). Interim assessments were performed at 4, 8, 12 and 16 weeks and post-treatment at 24 weeks (additional secondary outcome).
Time Frame: 20 weeks
Population: Estimation done using mixed-model ANOVA which includes all available data from all time points for all subjects. This analysis reduces bias compared to an analysis at each time point that excludes subjects with missing data. All study subjects were included, even if they did not have data observed at the given time point. In addition to missing data shown in Participant Flow table, outcome-specific missing data for 1 additional Arm A subject at week 12.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 15 | 15
score on a scale | 3.50 [2.59 to 4.40] | 3.55 [2.75 to 4.36]
Statistical Analysis 1: Comparison: Arm A vs Arm B; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.910, Mixed Models Analysis — A two-sided 5% significance level was used for all tests without multiplicity adjustment between multiple endpoints; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.06, 95% CI 2-sided [-1.13 to 1.01] — For difference calculation, Arm A - Arm B

6. Secondary Outcome: Jaw Function Limitation Scale (JFLS-8) at 20 Weeks
Description: Jaw Function Limitation Scale (JFLS-8) at 20 weeks: 0 (Better) - 10 (Worse).Interim assessments were performed at 4, 8, 12 and 16 weeks and post-treatment at 24 weeks (additional secondary outcome).
Time Frame: 20 weeks
Population: as for outcome 4
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 15 | 15
score on a scale | 0.47 [-0.22 to 1.16] | 0.48 [-0.14 to 1.11]
Statistical Analysis 1: Comparison: Arm A vs Arm B; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.972, Mixed Models Analysis — A two-sided 5% significance level was used for all tests without multiplicity adjustment between multiple endpoints; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.01, 95% CI 2-sided [-0.83 to 0.80] — For difference calculation, Arm A - Arm B

7. Secondary Outcome: Patient Health Questionnaire (PHQ-4) at 20 Weeks
Description: Depressive and Anxiety symptoms using Patient Health Questionnaire (PHQ-4) at 20 weeks: 0 (Better) - 12 (Worse). Interim assessments were performed at 4, 8, 12 and 16 weeks and post-treatment at 24 weeks (additional secondary outcome).
Time Frame: 20 weeks
Population: Estimation done using mixed-model ANOVA which includes all available data from all time points for all subjects. This analysis reduces bias compared to an analysis at each time point that excludes subjects with missing data. All study subjects were included, even if they did not have data observed at the given time point. In addition to missing data shown in Participant Flow table, outcome-specific missing data for 1 additional Arm A subject at week 12, 1 Arm B at week 4, and 1 Arm B at week 8.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 15 | 15
score on a scale | 4.42 [2.40 to 6.45] | 1.62 [-0.29 to 3.53]
Statistical Analysis 1: Comparison: Arm A vs Arm B; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.037, Mixed Models Analysis — A two-sided 5% significance level was used for all tests without multiplicity adjustment between multiple endpoints; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 2.81, 95% CI 2-sided [0.18 to 5.43] — For difference calculation, Arm A - Arm B

8. Secondary Outcome: Somatic Symptoms Scale (SSS-8) at 20 Weeks
Description: Assessment of somatic symptoms using the Somatic Symptoms Scale (SSS-8) at 20 weeks: 0 (Better) - 32 (Worse). Interim assessments were performed at 4, 8, 12 and 16 weeks and post-treatment at 24 weeks (additional secondary outcome).
Time Frame: 20 weeks
Population: as for outcome 5
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 15 | 15
score on a scale | 6.46 [3.34 to 9.57] | 6.72 [3.86 to 9.57]
Statistical Analysis 1: Comparison: Arm A vs Arm B; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.885, Mixed Models Analysis — A two-sided 5% significance level was used for all tests without multiplicity adjustment between multiple endpoints; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.26, 95% CI 2-sided [-3.95 to 3.43] — For difference calculation, Arm A - Arm B

9. Secondary Outcome: Brief Pain Inventory (BPI) Pain Severity at 24 Weeks
Description: Assessment of pain severity using the Brief Pain Inventory (BPI) 4-item pain severity scale at 24 weeks: 0 (Better) - 10 (Worse). Interim assessments were performed at 4, 8, 12 and 16 weeks and end of treatment at 20 weeks (primary outcome).
Time Frame: 24 weeks.
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 15 | 15
score on a scale | 1.99 [0.89 to 3.09] | 1.51 [0.47 to 2.56]
Statistical Analysis 1: Comparison: Arm A vs Arm B; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.474, Mixed Models Analysis — A two-sided 5% significance level was used for all tests without multiplicity adjustment between multiple endpoints; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.47, 95% CI 2-sided [-0.87 to 1.81] — For difference calculation, Arm A - Arm B

10. Secondary Outcome: Brief Pain Inventory (BPI) Pain Interference at 24 Weeks
Description: Assessment of pain interference using the Brief Pain Inventory (BPI) 7-item pain intensity scale at 24 weeks: 0 (Better) - 10 (Worse). Interim assessments were performed at 4, 8, 12 and 16 weeks and end of treatment at 20 weeks (additional secondary outcome).
Time Frame: 24 weeks
Population: Estimation done using mixed-model ANOVA which includes all available data from all time points for all subjects. This analysis reduces bias compared to an analysis at each time point that excludes subjects with missing data. All study subjects were included, even if they did not have data observed at the given time point. In addition to missing data shown in Participant Flow table, outcome-specific missing data for 1 additional Arm A subject at week 12 and 1 additional Arm B subject at week 20.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 15 | 15
score on a scale | 1.23 [-0.08 to 2.54] | 1.42 [0.19 to 2.65]
Statistical Analysis 1: Comparison: Arm A vs Arm B; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.822, Mixed Models Analysis — A two-sided 5% significance level was used for all tests without multiplicity adjustment between multiple endpoints; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.19, 95% CI 2-sided [-1.94 to 1.56] — For difference calculation, Arm A - Arm B

11. Secondary Outcome: Average Daily Reported Pain Scores at 24 Weeks
Description: Assessment of pain using average of daily reported pain scores at 24 weeks; average of daily reported scores from days > week 20 and <= week 24. Pain scale: 0 (Better) - 10 (Worse). Interim assessments were performed at 4, 8, 12 and 16 weeks and end of treatment at 20 weeks (additional secondary outcome).
Time Frame: 24 weeks
Population: as for outcome 3
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 15 | 15
score on a scale | 2.01 [0.84 to 3.17] | 1.49 [0.41 to 2.58]
Statistical Analysis 1: Comparison: Arm A vs Arm B; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.455, Mixed Models Analysis — A two-sided 5% significance level was used for all tests without multiplicity adjustment between multiple endpoints; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.51, 95% CI 2-sided [-0.88 to 1.91] — For difference calculation, Arm A - Arm B

12. Secondary Outcome: % of Days Taking Medication for Pain at 24 Weeks
Description: Assessment of pain using the % of days taking medication for pain at 24 weeks; percentage of days calculated from days > week 20 and <= week 24. Interim assessments were performed at 4, 8, 12 and 16 weeks and end of treatment at 20 weeks (additional secondary outcome).
Time Frame: 24 weeks
Population: as for outcome 4
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage of days
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 15 | 15
percentage of days | 13.7 [-5.2 to 32.6] | 6.6 [-10.2 to 23.5]
Statistical Analysis 1: Comparison: Arm A vs Arm B; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.467, Mixed Models Analysis — A two-sided 5% significance level was used for all tests without multiplicity adjustment between multiple endpoints; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 7.1, 95% CI 2-sided [-12.8 to 27.0] — For difference calculation, Arm A - Arm B

13. Secondary Outcome: Pain Improvement Using the Patient Global Impression of Change in Pain at 24 Weeks
Description: Assessment of pain improvement using the patient global impression of change in pain scale at 24 weeks: 1 (Better) - 7 (Worse). Interim assessments were performed at 4, 8, 12 and 16 weeks and end of treatment at 20 weeks (additional secondary outcome).
Time Frame: 24 weeks
Population: as for outcome 5
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 15 | 15
score on a scale | 3.70 [2.89 to 4.52] | 3.56 [2.83 to 4.29]
Statistical Analysis 1: Comparison: Arm A vs Arm B; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.755, Mixed Models Analysis — A two-sided 5% significance level was used for all tests without multiplicity adjustment between multiple endpoints; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.14, 95% CI 2-sided [-0.79 to 1.07] — For difference calculation, Arm A - Arm B

14. Secondary Outcome: Jaw Function Limitation Scale (JFLS-8) at 24 Weeks
Description: Jaw Function Limitation Scale (JFLS-8) at 24 weeks: 0 (Better) - 10 (Worse).Interim assessments were performed at 4, 8, 12 and 16 weeks and end of treatment at 20 weeks (additional secondary outcome).
Time Frame: 24 weeks
Population: as for outcome 4
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 15 | 15
score on a scale | 0.92 [0.18 to 1.66] | 1.16 [0.45 to 1.87]
Statistical Analysis 1: Comparison: Arm A vs Arm B; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.613, Mixed Models Analysis — A two-sided 5% significance level was used for all tests without multiplicity adjustment between multiple endpoints; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.23, 95% CI 2-sided [-1.18 to 0.71] — For difference calculation, Arm A - Arm B

15. Secondary Outcome: Patient Health Questionnaire (PHQ-4) at 24 Weeks
Description: Depressive and Anxiety symptoms using Patient Health Questionnaire (PHQ-4) at 24 weeks: 0 (Better) - 12 (Worse). Interim assessments were performed at 4, 8, 12 and 16 weeks and end of treatment at 20 weeks (additional secondary outcome).
Time Frame: 24 weeks
Population: as for outcome 7
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 15 | 15
score on a scale | 3.58 [2.21 to 4.95] | 1.00 [-0.31 to 2.31]
Statistical Analysis 1: Comparison: Arm A vs Arm B; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.003, Mixed Models Analysis — A two-sided 5% significance level was used for all tests without multiplicity adjustment between multiple endpoints; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 2.58, 95% CI 2-sided [0.94 to 4.22] — For difference calculation, Arm A - Arm B

16. Secondary Outcome: Somatic Symptoms Scale (SSS-8) at 24 Weeks
Description: Assessment of somatic symptoms using the Somatic Symptoms Scale (SSS-8) at 24 weeks: 0 (Better) - 32 (Worse). Interim assessments were performed at 4, 8, 12 and 16 weeks and end of treatment at 20 weeks (additional secondary outcome).
Time Frame: 24 weeks
Population: as for outcome 5
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 15 | 15
score on a scale | 6.70 [3.46 to 9.94] | 5.51 [2.53 to 8.48]
Statistical Analysis 1: Comparison: Arm A vs Arm B; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.536, Mixed Models Analysis — A two-sided 5% significance level was used for all tests without multiplicity adjustment between multiple endpoints; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 1.19, 95% CI 2-sided [-2.70 to 5.08] — For difference calculation, Arm A - Arm B

ADVERSE EVENTS:
Time Frame: 24 weeks
Description: Subjects were questioned regarding any general health or oral complaints and symptoms they had experienced during each visit. Any findings were documented on the AE CRF. All AEs, regardless of severity or relationship to the treatments, were recorded. In addition, other important medical events that were deemed clinically important/serious based on PI judgement were recorded as AEs.
Arm/Group | Arm A | Arm B
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 9/15 | 7/15
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (N=15) | Arm B (N=15)
Constipation (Gastrointestinal disorders) | 1 (2) | 0 (0)
Wart (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Wart on the right leg below kneecap
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Discomfort on back of the neck after injection
Allergic reaction (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Allergic reaction late onset at the injection sites(Itching and Swelling-both Thighs)
Bruise (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Bruises on the left thigh
Facial pain (Nervous system disorders) | 0 (0) | 1 (1) — Facial pain after exam
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Itching (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) — Itching at injection site
Food poisoning (Gastrointestinal disorders) | 1 (1) | 1 (1)
Burning Sensation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — Burning Sensation at injection site
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) — Erythema at injection site
COVID-19 (Infections and infestations) | 2 (2) | 2 (2)
Sinus Headache (General disorders) | 0 (0) | 1 (1)
TMJ Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — TMJ Pain (Bilateral Arthralgia)
Myofascial Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — Bilateral Myofascial pain
Common cold (Infections and infestations) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (3) | 0 (0)
Drowsiness (General disorders) | 1 (1) | 0 (0)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Wrist sprain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Wrist sprain right hand due to fall
Ear infection (Ear and labyrinth disorders) | 0 (0) | 1 (1) — Left ear infection from foreign object injury
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Dislocated Shoulder (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — Dislocated Right Shoulder
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Sore throat (Infections and infestations) | 0 (0) | 1 (1)
Low grade fever (General disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-01-12): https://cdn.clinicaltrials.gov/large-docs/63/NCT04884763/Prot_SAP_000.pdf
  • Informed Consent Form (2023-08-10): https://cdn.clinicaltrials.gov/large-docs/63/NCT04884763/ICF_001.pdf